CLINICAL TRIAL: NCT03957135
Title: Multicenter Prospective Randomized Controlled Clinical Trial for Comparison Between Laparoscopic and Open Distal Pancreatectomy for Ductal Adenocarcinoma of the Pancreatic Body and Tail
Brief Title: Laparoscopic Versus Open Distal Pancreatectomy for Pancreatic Cancer: a Multicenter Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Severance Hospital (Other); Asan Medical Center (Other); Seoul St. Mary's Hospital (Other); Samsung Medical Center (Other); Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ho-Seong Han, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH-GS-HBP4
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Pancreas Neoplasm Malignant Resectable
Keywords: pancreas neoplasms; pancreatectomy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic distal pancreatectomy (Experimental): Patients receiving laparoscopic distal pancreatectomy for pancreatic tail and body cancer
  Interventions: Procedure: Laparoscopic distal pancreatectomy
- open distal pancreatectomy (Active Comparator): Patients receiving open distal pancreatectomy for pancreatic tail and body cancer
  Interventions: Procedure: open distal pancreatectomy

INTERVENTIONS:
Procedure: Laparoscopic distal pancreatectomy — Laparoscopic resection of the diseased portion of the pancreas for treatment of pancreatic cancer
  Arms: Laparoscopic distal pancreatectomy
Procedure: open distal pancreatectomy — Open resection of the diseased portion of the pancreas for treatment of pancreatic cancer
  Arms: open distal pancreatectomy

SUMMARY:
When pancreatic cancer of the body and tail is diagnosed, a distal pancreatectomy is planned. This operation can be performed with open surgery, or with laparoscopic surgery. This study is a multicenter randomized controlled trial to evaluate the operative outcomes and survival of open versus laparoscopic distal pancreatectomy for pancreatic cancer of the body and tail.

DETAILED DESCRIPTION:
* Purpose

To compare the safety and oncologic feasibility of open versus laparoscopic distal pancreatectomy for the treatment of pancreatic ductal adenocarcinoma (PDAC) of the body and tail.

* Study method

Multicenter prospective randomized controlled trial Noninferiority analysis Patients diagnosed with PDAC of the body and tail, without evidence of distant metastasis or direct invasion of adjacent organs, will be randomly allocated to either the open distal pancreatectomy group or the laparoscopic distal pancreatectomy group. Postoperative outcomes and survival data will be analyzed.

* Number of subjects

Sample size was calculated based on 2 year survival after pancreatectomy.

pA: 2 year survival of open distal pancreatectomy pB: 2 year survival of laparoscopic distal pancreatectomy

Null hypothesis: The 2 year survival of laparoscopic distal pancreatectomy is inferior to that of open distal pancreatectomy. H0: pA-pB≥δ

Alternative hypothesis: The 2 year survival of laparoscopic distal pancreatectomy is not inferior to that of open distal pancreatectomy. H1: pA-pB<δ

2 year survival of pancreatectomy (Shin et al, 2015) is 55.9% for open and 64.3% for laparoscopic distal pancreatectomy.

When α=5%, 1-β=80%, δ=10%, and one-sided analysis is performed with a power of 80%, the required number of subjects is 111 for each group.

With a drop rate of 10%, the final number of each group is 122, with a total of 244.

* Primary and Secondary endpoints

Primary endpoint: 2 year overall survival

Secondary endpoint: R0 resection rate, 2 year disease free survival, 2 year recurrence rate, complication rate, postoperative hospital stay, operative time, estimated blood loss

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance score 0-2
* Pancreatic ductal adenocarcinoma that is pathologically confirmed or shows characteristic radiologic features
* Patients with resectable pancreatic cancer at the time of surgery (Including borderline resectable pancreatic cancer at the time of diagnosis or Locally advanced pancreatic cancer after chemotherapy or radiation therapy)
* Lesion (within pancreatic body and tail) is located to the left of the left branch of the hepatic portal vein
* No remote metastasis in preoperative imaging and not adjacent to the superior mesenteric vein, superior mesenteric artery, and abdominal artery
* Patients without invasion of adjacent organs other than the left adrenal gland and mesocolon
* Patients with informed consent

Exclusion Criteria:

* Patients with remote metastasis at the time of diagnosis of pancreatic cancer
* History of other malignancy (Inclusive if there is no evidence of recurrence after 5 years of treatment)
* In the case of invasion of other organs other than the left adrenal gland and mesocolon
* Where major vascular resection, such as the portal vein or abdominal artery, is required to secure negative resection
* Recurrent pancreatic cancer
* Patients with underlying diseases at high risk of general anesthesia
* Preperitoneal or other organ metastases found during surgery
* In case of previously undergone pancreatic resection
* Other subject whom the investigator deems inappropriate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
2 year survival | 2 years
  Overall survival at 2 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Seong Han, M.D. Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Kyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoon YS, Lee KH, Han HS, Cho JY, Jang JY, Kim SW, Lee WJ, Kang CM, Park SJ, Han SS, Ahn YJ, Yu HC, Choi IS. Effects of laparoscopic versus open surgery on splenic vessel patency after spleen and splenic vessel-preserving distal pancreatectomy: a retrospective multicenter study. Surg Endosc. 2015 Mar;29(3):583-8. doi: 10.1007/s00464-014-3701-9. Epub 2014 Jul 9. PMID 25005018
- [Background] Yoon YS, Lee KH, Han HS, Cho JY, Ahn KS. Patency of splenic vessels after laparoscopic spleen and splenic vessel-preserving distal pancreatectomy. Br J Surg. 2009 Jun;96(6):633-40. doi: 10.1002/bjs.6609. PMID 19434700
- [Background] Shin SH, Kim SC, Song KB, Hwang DW, Lee JH, Lee D, Lee JW, Jun E, Park KM, Lee YJ. A comparative study of laparoscopic vs. open distal pancreatectomy for left-sided ductal adenocarcinoma: a propensity score-matched analysis. J Am Coll Surg. 2015 Feb;220(2):177-85. doi: 10.1016/j.jamcollsurg.2014.10.014. Epub 2014 Oct 31. PMID 25529901